CLINICAL TRIAL: NCT05513651
Title: Establishment of a Model for Predicting the Prognosis of HBV-related Decompensated Liver Cirrhosis Based on RFH-NPT
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-023
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-12

CONDITIONS: Liver Cirrhosis; Malnutrition
Keywords: prediction; malnutrition; cirrhosis; prognosis
MeSH Terms: conditions — Liver Cirrhosis; Malnutrition; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For all countries, chronic liver disease and liver cirrhosis is one of the important disease burdens. Malnutrition is an important complication of liver cirrhosis, which always runs through the course of liver cirrhosis. According to a lot of scientific research evidence, as the consensus of experts all over the world, malnutrition in patients with liver cirrhosis is closely related to poor outcome. Therefore, early and accurate identification of the risk of malnutrition is very important to improve the prognosis of patients with liver cirrhosis.

The purpose of this study was to study the relationship between malnutrition-related indexes and prognosis in patients with liver cirrhosis. 2000 patients with liver cirrhosis were prospectively included, laboratory indexes related to malnutrition and other evaluation indexes were recorded, and long-term follow-up was made to observe the short-term and long-term prognosis of patients with liver cirrhosis. At the same time, a prognostic prediction model was established based on multivariate Cox regression, and a series of in-depth studies and verification were carried out on this basis.

DETAILED DESCRIPTION:
Malnutrition is one of the most common complications associated with liver cirrhosis, which is more likely to occur in patients with decompensated liver cirrhosis. Malnutrition will further lead to muscle loss, that is, the occurrence of myomyositis, which is an important cause of adverse outcome in patients with liver cirrhosis. it is associated with increased risk of death, portal hypertension-related complications, increased infection rates and longer hospital stays. At the same time, liver cirrhosis with portal hypertension leads to esophageal and gastric varices and intestinal mucosal edema, which affects the function of the digestive system and poses a greater challenge to the nutritional maintenance of patients with liver cirrhosis. Therefore, timely nutritional assessment and early intervention decision-making on admission is an important aspect of clinical management of patients with liver cirrhosis.

For the screening of malnutrition in patients with liver cirrhosis, the commonly used screening tools are MST, MUST, NRS-2002, RFH-NPT and so on. For the screened high-risk population, further specific nutritional assessment is needed, there are four main types. The first is a diet-related assessment conducted by a professional dietitian. The second is the body composition analysis represented by muscle mass, such as bioelectrical impedance analysis (BIA), CT, ultrasound and so on. The third is the functional evaluation, of which the more common are five-meter walking speed and grip strength test. The fourth is part of the comprehensive evaluation tools, represented by SGA and RFH-SGA.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with liver cirrhosis

Exclusion Criteria:

* Patients who refuse the follow-up of outpatient department

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with liver cirrhosis were recruited. In addition, healthy volunteers who had normal liver function and normal BMI were recruited and acted as controls.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | up to 10 years
  All-cause mortality is death caused by any cause.
Liver-related mortality | up to 10 years
  Liver-related mortality refers to death from any liver-related disease, such as liver cirrhosis, liver cancer and other related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu C, Wu Y, Zhao F, Wang R, Zang Q, Jiao Z, Zhu Y, Yan T, Du J, Zhu L, Li W, Li Y, Fan Q, Wu A, Liu X, Liu D, Tang X, Xu X, Liao H, Li Y, Zhao Y, He Y, Yang Y. An RFH-NPT-based nomogram for predicting the long-term survival of liver cirrhosis patients: a multicenter study. Eur J Clin Nutr. 2026 Jan;80(1):87-95. doi: 10.1038/s41430-025-01648-4. Epub 2025 Jul 29. PMID 40731156